CLINICAL TRIAL: NCT00024232
Title: Pilot Trial of Humanized Monoclonal Antibody J591 in Patients With Progressive Androgen-Independent Prostate Cancer
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MSKCC-01030; CDR0000068903 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-2013
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Biological: monoclonal antibody huJ591

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of monoclonal antibody therapy in treating patients who have prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor effects of monoclonal antibody huJ591 in patients with progressive androgen-independent prostate cancer.
* Determine the biodistribution and dosimetry of this antibody in these patients.
* Determine the effect on biodistribution of the delivery sequence of unlabeled vs indium In 111-labeled antibody in these patients.
* Determine the HAHA response in patients treated with this regimen.
* Correlate the dose of monoclonal antibody huJ591 with antibody-dependent cellular cytotoxicity in these patients.

OUTLINE: Patients are assigned to one of two treatment groups.

* Group I: Patients receive monoclonal antibody huJ591 IV followed by indium In 111 monoclonal antibody huJ591 on day 1.
* Group II: Patients receive monoclonal antibody huJ591 concurrently with indium In 111 monoclonal antibody huJ591 as in group I.

Treatment in both groups repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for 4 weeks and then monthly for 3 months.

PROJECTED ACCRUAL: A total of 14 patients (7 per treatment group) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer
* Disease progression after prior castration

  * At least 3 rising PSA levels at least 1 week apart OR 2 rising levels at least 4 weeks apart
* New osseous lesions on bone scan and/or more than 25% increase in bidimensionally measurable soft tissue disease or appearance of new sites of disease by CT scan or MRI
* Testosterone no greater than 50 ng/mL

  * Medical therapy (e.g., gonadotropin-releasing hormone analogues) to maintain castrate level of testosterone should continue in the absence of surgical orchiectomy
* Progression of disease after discontinuation of prior anti-androgen therapy
* No requirement for palliative therapy within the past 12 weeks
* No active CNS or epidural primary tumor OR active CNS or epidural metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,500/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* Gamma-glutamyl-transferase less than upper limit of normal (ULN)
* AST less than ULN
* PT less than 14 seconds
* No prior autoimmune hepatitis

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No clinically significant cardiac disease (New York Heart Association class III or IV)

Pulmonary:

* No severe debilitating pulmonary disease

Other:

* Fertile patients must use effective contraception
* No active uncontrolled infection or infection requiring IV antibiotics
* No prior autoimmune disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior murine protein for diagnostic or therapeutic purposes
* No other concurrent anticancer immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered
* No concurrent anticancer chemotherapy

Endocrine therapy:

* See Disease Characteristics
* No concurrent anticancer hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* Concurrent radiotherapy to localized sites of disease (e.g., bone) allowed if the site does not contain sole measurable lesion

Surgery:

* See Disease Characteristics
* No concurrent surgery

Other:

* Recovered from all prior therapy
* At least 4 weeks since prior therapeutic investigational anticancer drugs
* At least 4 weeks since prior participation in therapeutic clinical trial with an experimental drug
* No prior diagnostic ProstaScint, Myoscint, or Oncoscint scans
* No other concurrent therapeutic investigational anticancer agents
* No concurrent participation in other therapeutic clinical trial with an experimental drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States